CLINICAL TRIAL: NCT02067221
Title: Comparison of Surgical Outcomes in the Treatment of Renal Stones Larger Than 1 Centimeters Between MPCNL and RIRS: a Single-center, Randomized, Prospective Study
Brief Title: Comparison of Surgical Outcomes Between MPCNL and RIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SK Telecom Consortium (Other)
Responsible Party: Principal Investigator, Hyeon Jeong, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPCNL Study
Record Dates: First submitted 2014-02-12; First posted 2014-02-20 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Renal Stone
Keywords: percutaneous nephrolithotomy; renal calculi; ureteroscopy
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIRS (retrograde intrarenal surgery) (Active Comparator): Use of flexible ureteroscopy to access and remove renal stones without percutaneous nephrostomy tract
  Interventions: Device: RIRS
- MPCNL (mini-perc) (Experimental): A new technique that reduced the size of percutaneous tract to make renal stone into small pieces.
  Patients will be randomized and assigned to each group at the ratio 1:1
  Interventions: Device: MPCNL

INTERVENTIONS:
Device: RIRS — * RIRS arm
  * Use of flexible ureteroscopy to access and remove renal stones without percutaneous nephrostomy tract
  Other Names: retrograde intrerenal surgery
  Arms: RIRS (retrograde intrarenal surgery)
Device: MPCNL — * MPCNL arm
  * A new technique that reduced the size of percutaneous tract to make renal stone into small pieces.
  Other Names: minimally invasive percuntaneous nephrolithotomy; mini-perc
  Arms: MPCNL (mini-perc)

SUMMARY:
The objective of this research is to investigate the surgical outcomes of minimally invasive percutaneous nephrolithotomy(MPCNL) and retrograde intrarenal surgery (RIRS)for patients with renal stone larger than 1cm.

DETAILED DESCRIPTION:
It is pointed out that there is the disadvantage of conventional PCNL technique which showed dramatic decrease in Hb and renal damage even though it has some advantages of a short operation time and a high stone-free rate. MPCNL and RIRS has recently been considered as very efficacious methods.

ELIGIBILITY:
Inclusion Criteria:

* The person who has been diagnosed with renal stone larger than 1cm renal and who has been supposed to undergo MPCNL or RIRS.
* The person who signed up for participation and agree with intention of clinical test.

Exclusion Criteria:

* The patient whose medical record has been omitted from database.
* The patient who has an anatomical abnormality of urinary tract and/or metabolic illness
* The patient who do not agree with the intention of the clinical study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
stone-free rate | postoperative 1 month
  We will check the non-contrast CT scan at postoperative 1month when the patient visit the outpatient department. If the patient does not have any residual stone fragment, it will be reported to 'success.' Otherwise, we will measure the size of each stone of residual fragments.

SECONDARY OUTCOMES:
pain | postoperative 1 day
  Visual analogue scale will be measured: 0 (no pain) -> 10 (the most worst pain ever experienced)
hemoglobin drop | postoperative 1 day
  preoperative Hb level - Hb level of immediate postoperative 1 day
occurrence of complications | postoperative 1 day, and the postop 1month at OPD
  occurrence of stricture in non-contrast CT scan history taking of hematuria or fever
hospital stay | postoperative 1 month
  calculation of days of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Cho, Ph.D, Study Director — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, South Korea